CLINICAL TRIAL: NCT00923520
Title: A Phase 1, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of Intravenous Dimethane Sulfonate (DMS612, NSC 281612) in Advanced Malignancies
Brief Title: A Phase 1, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous Dimethane Sulfonate (DMS612) in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090111; 09-C-0111; NCT00888121 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12-03

CONDITIONS: Renal Cell Carcinoma; Breast Cancer; Colon Cancer; Lung Cancer; Non-Hodgkin Lymphoma
Keywords: Solid Tumors; Phase I; Lymphoma; Dimethane Sulfonate (DMS612, NSC 281612); Cancer; Solid Tumor; Renal Cell Cancer; Kidney Cancer; Breast Cancer; Colon Cancer; Lung Disease; Non-Hodgkin Lymphoma; NHL
MeSH Terms: conditions — Carcinoma, Renal Cell; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms; Kidney Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- 1 (Experimental): DMS 612 on day 1 and 2 with doses starting at 3.5mg/m2 to 18.5mg/m2 every 21 days until MTD is reached
  Interventions: Drug: DMS 612

INTERVENTIONS:
Drug: DMS 612 — DMS 612 on day 1 and 2 with doses starting at 3.5mg/m2 to 18.5mg/m2 every 21 days until MTD is reached

SUMMARY:
Background:

* Dimethane sulfonate (DMS612) is an investigational drug that is being administered to humans for the first time in people with advanced tumors. More information on the maximum tolerated dose of DMS612 will help researchers identify whether the drug is suitable for use in treating certain kinds of cancer, particularly renal cell carcinoma.

Objectives:

* To determine the maximum tolerated dose of DMS612 (the highest dose that does not cause unacceptable side effects) and evaluate any side effects.
* To see if DMS612 has any effect on patients tumors through blood tests and laboratory studies.
* To learn how the body processes DMS612.

Eligibility:

* Patients 18 years of age and older who have been diagnosed with cancer that has not responded well to standard treatments.

Design:

* Pre-treatment evaluation visit to determine eligibility:
* Physical examination
* Blood and urine tests
* Chest X-ray; electrocardiogram; CAT scan of chest, abdomen, pelvis, and other areas of the body if needed
* Other possible tests, such as magnetic resonance imaging (MRI) or positron emission tomography (PET)
* Patients will receive one dose of DMS612 by intravenous infusion once a week for 3 weeks, followed by 1 week without the drug. Doses will be adjusted based on possible side effects and cancer response. The disease will be evaluated after three cycles of the drug.
* Evaluations during the treatment period:
* Physical examination and reviews of side effects.
* Blood draws to evaluate the effectiveness of the drug, and how it is processed by the body.
* CAT scan at the end of every two cycles (every 8 weeks).
* Other scans and imaging procedures as required by the study doctors.

DETAILED DESCRIPTION:
Background:

* The dimethane sulfonates are a group of agents that were identified as active against renal cell carcinoma in the NCI anticancer drug screen.
* In vitro studies showed that dimethane sulfonates have properties in common with alkylating agents, but are unlike conventional alkylators (such as nitrogen mustards, BCNU, or busulfan) in that they are active against renal cell carcinoma (RCC).

Objective:

Primary:

-To determine dose-limiting toxicity (DLT), MTD and recommended phase II dose (RPTD) of dimethane sulfonate (DMS612, NSC 281612) when administered by intravenous (IV) bolus on day 1 and 2 of a 21-day cycle.

Eligibility:

* Patients must have histologically confirmed solid tumor malignancy or lymphoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Any prior chemotherapy therapy is allowed in this protocol. No more than 2 prior cytotoxic chemotherapy regimens are allowed.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of Dimethane sulfonate in patients less than 18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* ECOG performance status 0-2 (Karnofsky greater than or equal to 60%,).
* Life expectancy of 3 months or greater.
* Patients must have acceptable organ and marrow function as defined below: leukocytes greater than or equal to 3,000/mcL, absolute neutrophil count greater than or equal to 1,500/mm(3), platelets greater than or equal to 100,000/, mm(3) total bilirubin within normal institutional limits, AST(SGOT)/ALT(SGPT), less than or equal to 2.5 times the institutional upper limit of normal, creatinine within normal institutional limits or creatinine clearance greater than 50mL/min for patients with creatinine levels above institutional normal.

Design:

This is a Phase I study of the safety, pharmacokinetics, pharmacodynamics and antitumor activity of IV DMS612, NSC 281612, designed as an open-label, dose-escalation study to determine the RPTD of DMS612, NSC 281612 based on safety and pharmacokinetics. With the 02/09/2015 amendment and change in schedule to evaluate a day 1 and 2 dosing every 6 weeks the following schema will be used:

Dose Level Dose of NSC 281612 Escalation (%)

* 1 3.5 mg/m2 on Day 1 and 2 -33

  4A 4.5 mg/m2 on Day 1 and 2 ---

  5A 6 mg/m2 on Day 1 and 2 33

  6A 8 mg/m2 on Day 1 and 2 67

  7A 10.5 mg/m2 on Day 1 and 2 33

  7B 10.5 mg/m2 on Day 1 and 2 q 6 weeks ---

  8A 14 mg/m2 on Day 1 and 2 33

  8B 14 mg/m2 on Day 1 and 2 q 6 weeks --

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumor malignancy or lymphoma that is metastatic or unresectable and for which effective therapy does not exist or is no longer effective.
* Any prior chemotherapy therapy is allowed in this protocol. No more than 2 prior cytotoxic chemotherapy regimens are allowed for eligibility. Non-myelotoxic therapies such as sunitinib and sorafenib or everolimus are not considered "cytotoxic chemotherapies".Patients must be greater than or equal to 4 weeks from prior radiation or cytotoxic chemotherapy, except greater than or equal to 6 weeks for mitomycin C and nitrosoureas; greater than or equal to 2 weeks from hormonal therapy; greater than or equal to 4 weeks from prior experimental therapy; greater than or equal to 4 weeks from monoclonal antibody therapy (cetuximab, bevacizumab), greater than or equal to 2 weeks from sorafenib, sunitinib or temsirolimus and greater than or equal to 8 weeks from prior UCN01 treatment. Patients with prostate cancer may continue ongoing LHRH agonist therapy. Patients with bone metastases or hypercalcemia who began intravenous bisphosphonate treatment prior to study entry may continue this treatment.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of dimethane sulfonate in patients less than 18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* ECOG performance status 0-2 (Karnofsky greater than or equal to 60%,).
* Life expectancy of 3 months or greater.
* Patients must have acceptable organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mm(3)
  * absolute neutrophil count greater than or equal to 1,500/ mm(3)
  * platelets greater than or equal to 100,000/ mm(3)
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * 24 hour urine creatinine clearance greater than 50 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal (may use creatinine clearance Cockcroft-Gault Equation).
* The effects of dimethane sulfonate on the developing human fetus are unknown. For this reason and because alkylating agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least 3 months after study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Willing to comply with study procedures and follow-up.

EXCLUSION CRITERIA:

* Patients who have not recovered (CTC less than or equal to grade I) from adverse events due to prior treatments
* Patients may not have received more than 2 prior cytotoxic regimens.
* Patients may not be receiving any other investigational agent with therapeutic anticancer intent.
* Patients with history of CNS metastasis, unless control has been achieved with either radiation or surgical resection at least 3 months prior to enrollment on study.
* Patients who have had radiation to the pelvis or other bone marrow-bearing sites will be considered on a case by case basis and may be excluded if the bone marrow reserve is not considered adequate (greater than 25% of bone marrow irradiated).
* Uncontrolled medical illness including, but not limited to, ongoing or active infection, chronic or acute hepatitis, renal failure, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because DMS612 is likely to have toxicities similar to the alklyating agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DMS612, breastfeeding should be discontinued if the mother is treated with DMS612.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with DMS612. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients are not eligible for the study if taking cytochrome P450-inducing anticonvulsants. This applies to patients with brain metastasis or those taking anticonvulsant for another reason (ie. Epilepsy).
* Patients diagnosed with alcoholism may not be treated with disulfiram.
* Patients may not be receiving agents thought to inhibit or induce the cytochrome p450 isoenzyme CYP3A4.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03-25; Primary Completion 2016-05-12 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose | End of Cycle 1
  Number of DLTs in on a given dose level.

SECONDARY OUTCOMES:
Evaluate non-dose limiting toxicity | Treatment Completion
  Number of overall toxicities on the study.
PK | Collection of Samples
  Drug level in blood
Anti-tumor Effects | Disease Progression
  Proportion of patients whose tumors shrunk after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Bishop JB, Wassom JS. Toxicological review of busulfan (Myleran). Mutat Res. 1986 Jul;168(1):15-45. doi: 10.1016/0165-1110(86)90020-5. PMID 3713721
- [Background] Cangiano T, Liao J, Naitoh J, Dorey F, Figlin R, Belldegrun A. Sarcomatoid renal cell carcinoma: biologic behavior, prognosis, and response to combined surgical resection and immunotherapy. J Clin Oncol. 1999 Feb;17(2):523-8. doi: 10.1200/JCO.1999.17.2.523. PMID 10080595
- [Background] Escudier B, Pluzanska A, Koralewski P, Ravaud A, Bracarda S, Szczylik C, Chevreau C, Filipek M, Melichar B, Bajetta E, Gorbunova V, Bay JO, Bodrogi I, Jagiello-Gruszfeld A, Moore N; AVOREN Trial investigators. Bevacizumab plus interferon alfa-2a for treatment of metastatic renal cell carcinoma: a randomised, double-blind phase III trial. Lancet. 2007 Dec 22;370(9605):2103-11. doi: 10.1016/S0140-6736(07)61904-7. PMID 18156031